CLINICAL TRIAL: NCT01637233
Title: Maraviroc Switch Central Nervous System (CNS) Substudy: a Substudy of MARCH, a Randomised, Open-label Study to Evaluate the Efficacy and Safety of Maraviroc (MVC) as a Switch for Either Nucleoside or Nucleotide Analogue Reverse Transcriptase Inhibitors (N(t)RTI) or Boosted Protease Inhibitors (PI/r) in HIV-1 Infected Individuals With Stable, Well-controlled Plasma HIV-RNA While Taking Their First N(t)RTI + PI/r Regimen of Combination Antiretroviral Therapy (cART).
Brief Title: MARCH Central Nervous System Substudy
Status: Completed | Type: Observational
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: MARCH-Kirby CNS; 2011-002107-15 (EudraCT Number)
Record Dates: First submitted 2012-06-27; First posted 2012-07-11 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: HIV-1 Infection
Keywords: HIV-1 infection; neurocognitive function; switch study
MeSH Terms: interventions — Tenofovir; Emtricitabine; Zidovudine; Lamivudine; abacavir; Ritonavir; Lopinavir; Darunavir; Atazanavir Sulfate; fosamprenavir; Protease Inhibitors; Maraviroc

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and CSF
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- NRTI + PI: This is the randomisation of the main study, Arm 1
  Interventions: Drug: Arm 1 TNucleotide Analogue Reverse Transcriptase Inhibitors and Boosted Protease Inhibitors
- maraviroc + PI: this is the randomisation of the main study, Arm 2
  Interventions: Drug: Arm 2 Maraviroc and Protease Inhibitors
- maraviroc + NRTI: this is the randomisation of the main study, Arm 3
  Interventions: Drug: Arm 3 Maraviroc and Nucleotide Analogue Reverse Transcriptase Inhibitors

INTERVENTIONS:
Drug: Arm 1 TNucleotide Analogue Reverse Transcriptase Inhibitors and Boosted Protease Inhibitors — NRTI+PI
  Other Names: tenofovir; emtricitabine; zidovudine; lamivudine; abacavir; Ritonavir; lopinavir; darunavir; atazanavir; fosamprenavir
  Groups: NRTI + PI
Drug: Arm 2 Maraviroc and Protease Inhibitors — maraviroc + PI
  Other Names: maraviroc; Ritonavir; lopinavir; darunavir; atazanavir; fosamprenavir
  Groups: maraviroc + PI
Drug: Arm 3 Maraviroc and Nucleotide Analogue Reverse Transcriptase Inhibitors — maraviroc + NRTI
  Other Names: maraviroc; tenofovir; emtricitabine; zidovudine; lamivudine; abacavir
  Groups: maraviroc + NRTI

SUMMARY:
This substudy is a prospective, observational, open-label, randomised study within the MARCH study. The purpose of this substudy is to investigate the changes in cerebral function parameters at 5 timepoints over 96 weeks of the three different treatment arms within the MARCH study. The investigators hypothesise that there will be improvements in cerebral function in those patients randomised, as part of the parent study, into the maraviroc arms.

the assessments in this CNS substudy will include:

1. Neurocognitive function as assessed by a computerised testing battery called CogState;
2. changes in cerebral metabolites as measured via 1H Magnetic Resonance Spectroscopy (1H-MRS)

In those randomised to the maraviroc arms (arms 2 and 3) there is an optional Lumbar puncture at week 48. The cerebrospinal fluid will be used to measure maraviroc levels and an ultrasensitive CSF HIV-1 viral load. These results will be matched with levels in the plasma.

DETAILED DESCRIPTION:
this is detailed above, this is a substudy of MARCH

ELIGIBILITY:
Inclusion Criteria:

* Provision of written, informed consent for participation in the substudy
* Enrolled into the substudy either at or before the week 0 visit of the main study

Exclusion Criteria:

* Pre-existing CNS diseases
* Recent head injury (past three months)
* Current history of major depression or psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participants in the MARCH main study who are eligible for the CNS substudy and provide written informed consent for participation
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To assess changes in NC function over 96 weeks, measured via a computerised testing battery in HIV-infected subjects stable on antiretroviral therapy randomised to three different treatment approaches | 96 weeks
  using CogState testing at 5 timepoints, weeks 0, 12, 24, 48, 96
To assess changes in cerebral metabolites over 96 weeks, measured via 1H Magnetic Resonance Spectroscopy (1H-MRS), in HIV-infected subjects stable on antiretroviral therapy randomised to three different treatment approaches | 96 weeks
  Assessment of CNS metabolites via 1H-MRS at week 0, 48, 96
  * Cerebral metabolites in frontal white and grey voxels, and basal ganglia will be measured
  * Measurable metabolites will include assessment of neuronal markers, N-acetyl-aspartate, and inflammatory markers, myo-Inositols and Choline

SECONDARY OUTCOMES:
to assess CSF HIV-1 RNA and CSF maraviroc concentration (in the MVC treatment arms) versus plasma HIV -1 RNA and MVC concentration after 48 weeks of therapy | 48 weeks
  A LP examination at week 48 (optional and only in the MVC treatment arms, and only if there is no contraindication to LP) to assess, with matched plasma samples:
  * CSF MVC concentration
  * CSF HIV-1 RNA
  * CSF biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Alan Winston, MD, Principal Investigator — Imperial Healthcare, London, UK
Locations (6):
- Argentina (3):
  - Fundación IDEAA, Buenos Aires, Buenos Aires
  - Hospital Ramos Mejía, Buenos Aires
  - CAICI, Rosario
- Chulalongkorn University Hospital, Bangkok, Bangkok, Thailand
- United Kingdom (2):
  - Brighton & Sussex University NHS Trust, Brighton, Sussex
  - Imperial Healthcare, St. Mary's Hospital, London